CLINICAL TRIAL: NCT06245642
Title: A Multi-center, Randomized, Double-blind, Positive Parallel Control Study of Compound Ciwujia Granules in the Treatment of Chronic Fatigue Syndrome (Spleen-kidney Deficiency Syndrome, Heart-spleen Deficiency Syndrome)
Brief Title: Compound Ciwujia Granules Treat Chronic Fatigue Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heilongjiang Quanle Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FFCWJKE-RCT-002
Record Dates: First submitted 2024-01-24; First posted 2024-02-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive control group (Active Comparator): Guipi Granules + Compound Ciwujia Granules simulator
  Interventions: Drug: Compound Ciwujia Granules, Guipi Granules
- Experimental group (Experimental): Compound Ciwujia Granules + Guipi Granules simulator
  Interventions: Drug: Compound Ciwujia Granules, Guipi Granules

INTERVENTIONS:
Drug: Compound Ciwujia Granules, Guipi Granules — Experimental group: Basic treatment + Compound Ciwujia Granules + Guipi Granules simulator orally for 6 weeks; Positive drug control group: basic treatment + Guipi Granules + Compound Ciwujia Granules simulant orally for 6 weeks.
  Other Names: Primary therapy

SUMMARY:
To observe the improvement of Chalder scale score in patients with chronic fatigue syndrome treated by Compound Ciwujia Granules. Improvement =[(baseline score - post-treatment score)/baseline score]*100%

DETAILED DESCRIPTION:
After being informed of the study and potential risks, all subjects who have given informed consent undergo a 2-week screening period to determine eligibility, and on day 0, subjects who meet eligibility requirements will be randomly assigned in a double-blind way. The patients were treated with Compound Ciwujia Granules + Guipi Granules/placebo (experimental group) and Compound Ciwujia Granules/placebo + Guipi Granules (positive control group) at a ratio of 1:1 for 6 weeks. Compound Ciwujia Granules/placebo 8g per bag, 2 times a day, 1 bag each time, Guipi Granules, 3g per bag, taken with boiling water. 1 bag (3g) at a time, 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of Western medicine for chronic fatigue syndrome;
* Meet the diagnostic criteria of spleen and kidney deficiency syndrome or heart and spleen deficiency syndrome of traditional Chinese medicine;
* Chalder scale score greater than 12 points;
* Age 18-70 years old, gender is not limited;
* Agree to participate in this clinical study, voluntarily sign informed consent, and agree to participate in visits, examinations, and treatments according to the requirements of the research protocol.

Exclusion Criteria:

* Combined with mental disorders such as severe anxiety and severe depression;
* Secondary fatigue caused by drugs or other reasons;
* Patients with serious primary diseases such as cardiovascular and cerebrovascular, liver, kidney and hematopoietic system, malignant tumors, and other serious complications; Abnormal liver and kidney function ALT, AST≥ 1.5 times the upper limit of normal value, Cr > the upper limit of normal value;
* Women who are pregnant, breastfeeding or who may become pregnant in the study and cannot use effective contraception;
* Have received relevant treatment and may affect the observed effect indicators;
* Suspected to have a history of drug abuse or other patients who do not meet the eligibility criteria;
* Allergic physique and allergic to the drug;
* Uncontrolled hypertension (DBP > 100mmHg or SBP > 160 mmHg);
* Diabetic patients;
* Those that the researcher thinks are not suitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
The subjects' Chalder scale scores changed after 3 and 6 weeks of treatment | Screening/Baseline period (Week -2 to Day 0), Treatment period (Week 3 ± 5 days), Treatment period (Week 6 ± 5 days)
  Based on the results of a multicenter RCT on CFS conducted earlier, it was found that the higher the baseline Chalder scale score, the greater the decrease in the score after treatment. Therefore, to reduce the differences in efficacy caused by the baseline, we used the nimodipine efficacy calculation method to evaluate the improvement in Chalder scale scores.
  Calculation method: Improvement = [(Baseline score - Post-treatment score) / Baseline score] * 100%

SECONDARY OUTCOMES:
Changes in Chalder scale scores and sub-scores | Screening/Baseline period (Week -2 to Day 0), Treatment period (Week 3 ± 5 days), Treatment period (Week 6 ± 5 days)
Changes in TCM syndrome scores and sub-scores | Screening/Baseline period (Week -2 to Day 0), Treatment period (Week 3 ± 5 days), Treatment period (Week 6 ± 5 days)
Changes in scores of EQ-5D-5L Quality of Life questionnaire | Screening/Baseline period (Week -2 to Day 0), Treatment period (Week 3 ± 5 days), Treatment period (Week 6 ± 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotian Zhang, Master, Principal Investigator — Shanghai Shuguang Hospital, Shanghai University of Traditional Chinese Medicine; Weian Yuan, Doctor, Principal Investigator — Shanghai Shuguang Hospital, Shanghai University of Traditional Chinese Medicine
Locations (1):
- Shanghai Shuguang Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmes GP, Kaplan JE, Gantz NM, Komaroff AL, Schonberger LB, Straus SE, Jones JF, Dubois RE, Cunningham-Rundles C, Pahwa S, et al. Chronic fatigue syndrome: a working case definition. Ann Intern Med. 1988 Mar;108(3):387-9. doi: 10.7326/0003-4819-108-3-387. PMID 2829679
- [Background] Wu Qiao, Gao Jing, Bo Ding Xi, etc. Meta-analysis of prevalence of chronic fatigue syndrome in Chinese population [J]. Youjiang Med, 2019,48(10):727-735. (in Chinese) DOI:10.3969/j.issn.1003-1383.2020.10.002.
- [Background] Maher KJ, Klimas NG, Fletcher MA. Chronic fatigue syndrome is associated with diminished intracellular perforin. Clin Exp Immunol. 2005 Dec;142(3):505-11. doi: 10.1111/j.1365-2249.2005.02935.x. PMID 16297163
- [Background] Kang Meihua. Chronic fatigue syndrome [J]. International journal of pediatrics, 2011, 42 (5) : 516-518521. The DOI: 10.3760 / cma. J.i SSN. 1673-4408.2011.05.029.
- [Background] Qing · Yu Jing. Synopsis of Golden Chamber. Kuang Huitao, tidy up. Taiyuan: Shanxi Science and Technology Press, 2012:94-9. (in Chinese [6] Rong Haibo, Zhang Shiming. Professor Zhang Shiming Chinese medicine classification diagnostic criteria of exercise fatigue. Journal of Chengdu University of Traditional Chinese Medicine [J], 2017,40 (4):72.
- [Background] Man Shanshan, Bian Yuhong, Gu Zhimin, et al. Analysis of anti-fatigue mechanism of traditional Chinese medicine. Tianjin Pharmacy [J], 2014, 26(2):62-65. (in Chinese)
- [Background] Zhang Shan. Protective effect and mechanism of Acanthopanax injection on cardiotoxicity and cerebral ischemic injury [D]. Tianjin: Tianjin Medical University, 2019.
- [Background] Wang Bingzhu. Huangdi's internal channels [M]. Beijing: The Commercial Press, 1955:59
- [Background] Fukuda K,StrcdusS.HickieI,eta1．The chornic fatiyue syndrome:a comprehensive approach it，Sdenfinition and study[J]．Annal of internal Mendicine，1994,121：953-959．
- [Background] Luo Ren, Kuang Rijian, ZHAO Xiaoshan, Huang Jianhua, Clinical Guidelines for the treatment of chronic fatigue syndrome with new Chinese medicines [C]. Chinese Association of Chinese Medicine Sub-Health Branch General election and
- [Background] Yuan Wan-Li, KANG Ming-xiang, WU Zhi-Hui, YU Ping. Chronic fatigue syndrome of traditional Chinese medicine standard of clinical research [J]. Journal of shaanxi traditional Chinese medicine, 2009, 30 (5) : 515-517. The DOI: 10.3969 / j.i SSN. 1000-7369.2009.05.001.